CLINICAL TRIAL: NCT00971204
Title: Clinical Study of the CardioFocus Endoscopic Ablation System - Adaptive Contact (EAS-AC) for the Treatment of Symptomatic Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-2734
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation; PAF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with HeartLight System (Experimental): Treatment of paroxysmal atrial fibrillation (PAF) with HeartLight System
  Interventions: Device: CardioFocus HeartLight Endoscopic Ablation System

INTERVENTIONS:
Device: CardioFocus HeartLight Endoscopic Ablation System — PVI ablation

SUMMARY:
This is a demonstration of safety and efficacy of the ablation for pulmonary vein isolation in the treatment of paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years
* paroxysmal atrial fibrillation
* failure of at least one AAD
* others

Exclusion Criteria:

* overall good health as established by multiple criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burke Barret, Study Director — CardioFocus, Inc.
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pacific Heart Institute, Santa Monica, California
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mt. Sinai Hospital, New York, New York
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - University Of Virginia Health System, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment With EAS-AC: Treatment of PAF with EAS-AC
  CardioFocus Endoscopic Ablation System - Adaptive Contact (EAS-AC): PVI ablation
Period: Overall Study
Arm/Group | Treatment With EAS-AC
Started | 100 (100 enrolled participants)
Treated | 86
Completed | 76 (86 participants were treated and of these 86, 76 completed the study.)
Not Completed | 24
Not completed — Did not meet all criteria-not treated | 14
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Population: 100 participants were enrolled in the study. 86 participants that met all inclusion/exclusion criteria received treatment with the HeartLight System and are included in the reported results.
Groups:
- Treatment With HeartLight: Treatment of PAF with HeartLight System PVI ablation
Arm/Group | Treatment With HeartLight
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 79
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Recurrence of Atrial Fibrillation
Description: Absence of symptomatic atrial fibrillation lasting one minute or more beyond the 90-day blanking period during the 12 month evaluation period.
Time Frame: 12 months
Population: Primary Effectiveness Endpoint participants. Of the 86 enrolled and treated participants, 84 were evaluable for the effectiveness endpoint.
Measure: Number; unit: successful participants
Groups:
- Treatment With HeartLight: Treatment of PAF with HeartLight System
  CardioFocus HeartLight Endoscopic Ablation System: PVI ablation
Arm/Group | Treatment With HeartLight
Number analyzed (Participants) | 84
successful participants | 50

ADVERSE EVENTS:
Groups:
- Treatment With HeartLight: Treatment of PAF with HeartLight
Arm/Group | Treatment With HeartLight
Serious Adverse Events (participants affected / at risk) | 14/86
Other Adverse Events (participants affected / at risk) | 23/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With HeartLight (N=86)
Cardiac perforation, pericardial effusion, tamponade (Cardiac disorders) | 4 (4) — Participants may have more than one reported AE.
Pericarditis (Cardiac disorders) | 7 (7) — Participants may have more than one reported AE.
Phrenic nerve injury (Musculoskeletal and connective tissue disorders) | 5 (5) — Participants may have more than one reported AE.
Death, unrelated to investigational device (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With HeartLight (N=86)
Chest pain/discomfort (Cardiac disorders) | 10 (12)
Pericarditis (Cardiac disorders) | 8 (8)
Phrenic nerve injury (Musculoskeletal and connective tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No